CLINICAL TRIAL: NCT00041535
Title: A Phase I/II Randomized, Controlled Study of OGT 918 in Patients With Neuronopathic Gaucher Disease
Brief Title: OGT 918-006: A Phase I/II Randomized, Controlled Study of OGT 918 in Patients With Neuronopathic Gaucher Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 020243; 02-N-0243
Record Dates: First submitted 2002-07-09; First posted 2002-07-10 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-03-03

CONDITIONS: Gaucher Disease
Keywords: Eye Movements; Saccades; Metabolic; Lysosomal; Myoclonus; Gaucher Disease; Neuronopathic Gaucher Disease
MeSH Terms: conditions — Gaucher Disease; Myoclonus | interventions — miglustat

INTERVENTIONS:
Drug: OGT 918

SUMMARY:
Gaucher disease is an inherited functional deficiency of glucocerebrosidase. This enzyme breaks down a fatty substance (lipid) called glucocerebroside, which is present in all cells of the body. When cells renew themselves, the lipids must be broken down and discarded. Because the enzyme does not function well, the lipid builds up in certain tissues, such as the liver and spleen. The nervous system is involved as well; memory is impaired and it is difficult to move the eyes from side to side. It has been shown that repeated infusions of glucocerebrosidase help break down the stored lipid. However, this treatment does not improve any neurological symptoms.

A medicine called OGT 918 has been shown to slow the production of the lipid that builds up in Gaucher disease. It also has been shown to enter the brain. It is hoped that taking OGT 918 will reduce the storage of glycolipids in cells and improve the neurological symptoms of the disease. This clinical trial seeks to evaluate OGT 918 as a treatment for neuronopathic Gaucher disease by assessing changes in eye movement velocity. A secondary goal is to assess the clinical safety and tolerability of OGT 918 therapy.

Up to 30 patients from the National Institutes of Health and the Institute of Child Health (London) will be randomly assigned to OGT 918 or no treatment for 12 months. Study participants must be clinically diagnosed with neuronopathic Gaucher disease, 12 years of age or older, and able to swallow capsules. They must have been stable on ERT for at least 6 months before the study.

Patients receiving OGT 918 will receive a dose of 200 mg OGT 918 three times daily. Data analysis will be done after 12 months. The study will be extended up to 12 months to collect safety and efficacy data. All patients who complete the main study and enter the extension study will receive OGT 918.

During a 4-week screening period, eye movement velocity will be measured. These assessments will be repeated at months 12 and 24. Also at screening and months 12 and 24, the following tests will be done: MRI/CT, to measure spleen and liver volume; pulmonary imaging (by X-ray) and function tests; nerve conduction velocity studies and neuropsychological assessments; evoked response studies (to measure how the brain conducts electrical messages); and tremor measurements. Additional assessments for tremor will be conducted at months 6 and 18.

Plasma samples will be obtained every 3 months to measure disease markers and safety profiles. Proteasome samples will be taken at screening and month 6 to identify proteins that may be associated with Gaucher disease. Blood will be obtained at month 1 from the first 6 consenting patients who have been randomly assigned to take OGT 918. These patients will also have a cerebrospinal fluid sample taken by lumbar puncture at month 1. These samples will be measured for how much OGT 918 is present.

All patients receiving OGT 918 will have an initial assessment 1 week after beginning treatment to evaluate tolerance of the therapy. Clinic visits will be every 3 months. All patients will be asked to keep a simple diary of adverse events and dietary information. Dose levels may be reduced if a patient experiences severe gastrointestinal problems.

DETAILED DESCRIPTION:
Gaucher disease is an inherited functional deficiency of glucocerebrosidase (beta-glucosidase) which leads to glycolipid accumulation in various tissues. OGT 918 is a reversible inhibitor of glucosylceramide synthase, a key enzyme in the synthesis of glycolipids, and has shown beneficial effects in a clinical study in type 1 Gaucher disease.

The primary objective of this clinical trial is to evaluate OGT 918 as a treatment for neuronopathic Gaucher disease by assessing changes in saccadic eye movement velocity. Other markers of the disease will also be assessed, including neurological and pulmonary involvement. Secondary objectives are to assess the clinical safety and tolerability of OGT 918 therapy.

Up to 30 patients, recruited from the National Institutes Health, Bethesda, USA and the Institute of Child Health, London, U.K. will be randomized to OGT 918 or no treatment in a 2:1 ratio for the 12 month study period. Patients will be clinically diagnosed with neuronopathic Gaucher disease, 12 years of age or older, on a stable dose of enzyme replacement therapy (ERT) for at least 6 months and be able to swallow capsules. Randomization will be stratified based on whether or not the patient has undergone a splenectomy.

All patients will follow an identical visit schedule. Patients aged 12 years or over randomized to receive OGT 918 will commence treatment at a dose of 200 mg (2 x 100 mg capsules) OGT 918 three times daily. As some patients may experience initial gastrointestinal intolerance this dose may be modified, however the aim will be to maintain patients at the highest tolerable dose in order to achieve the most clinical benefit. Data analysis is planned, comparing OGT 918 to the no treatment group, when all patients have completed 12 months of the study. The study will be extended, up to a total of 12 additional months, to collect safety and efficacy data. The length of the extension study will be dependent on the results of the final analysis. All patients completing the main study, including those initially randomized to the no treatment group, will be able to participate in the extension study unless there are safety issues to prohibit this. All patients in the extension study will receive OGT 918.

Disease activity assessments will be conducted as indicated in the study flow charts. For a complete description of all study assessments, please refer to Section 7 of the main protocol. Where possible, study assessments will be blinded.

The effect of OGT 918 on the electro-oculographic characteristics of saccadic activity, specifically the amplitude/velocity characteristics (main sequence), will be the primary outcome variable. Saccadic velocity-amplitude relationship is decreased in neuronopathic Gaucher patients. This study will assess whether OGT 918 therapy is capable of improving or stopping any further deterioration of this ocular function.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with neuronopathic Gaucher disease, confirmed by clinical diagnosis, who if receiving enzyme replacement therapy have been stable on enzyme replacement therapy for at least 6 months or have successfully undergone a bone marrow transplant at least one year prior to study entry.

Patients who are at least 4 years old and can swallow a capsule.

EXCLUSION CRITERIA:

Patients younger than 18 years who are unable to give informed assent and/or whose legal guardian is unable to provide informed consent.

Patients aged 18 and over who cannot provide informed consent and/or whose legal guardian is unable to provide witnessed informed consent.

Fertile patients, who at the time of the study could be sexually active, and who do not agree to use adequate contraception throughout the study and for three months after cessation of OGT 918 treatment.

Patients who cannot tolerate the study procedures or who are unable to travel to the study center as required by this protocol.

Patients currently undergoing therapy with other investigational agents or patients taking drugs or food supplements which may interfere with gastrointestinal absorption or motility.

Patients suffering from clinically significant diarrhea (greater than 3 liquid stools per day for greater than 7 days) without definable cause within 3 months of the Screening Visit, or who have a history of significant gastrointestinal disorders.

Patients with an intercurrent medical condition that would render them unsuitable for the study e.g. HIV, hepatitis infection.

Patients who in the opinion of the investigator (for whatever reason) are thought to be unsuitable for the study.

Patients with an adjusted Creatinine Clearance of less than 70 ml/min/1.73m(2) (CrCl less than 70).

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2002-07-05; Study Completion 2007-03-21

CONTACTS AND LOCATIONS:
Locations (2):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States
- Institute of Child Health, London, United Kingdom

REFERENCES:
- [Background] Platt FM, Neises GR, Dwek RA, Butters TD. N-butyldeoxynojirimycin is a novel inhibitor of glycolipid biosynthesis. J Biol Chem. 1994 Mar 18;269(11):8362-5. PMID 8132559